CLINICAL TRIAL: NCT02693444
Title: Comparison of Strength and Constant Score Pre- and Post-Subacromial Injection for Full Thickness Rotator Cuff Tears
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low pool of subjects
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15081703
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Rotator Cuff; Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subacromial Lidocaine Injection (Active Comparator): Both of your shoulders will be examined and evaluated (shoulder survey). Following the exam, you will be randomized (assigned by chance, similar to a coin toss) to receive a 10cc (2 teaspoon) subacromial injection of lidocaine, will be given under ultrasound (using sound waves) guidance to your affected shoulder. A repeat shoulder exam will be performed and recorded
  Interventions: Drug: Lidocaine
- Subacromial Saline Injection (Placebo Comparator): Both of your shoulders will be examined and evaluated (shoulder survey). Following the exam, you will be randomized (assigned by chance, similar to a coin toss) to receive a 10cc (2 teaspoon) subacromial injection of saline, will be given under ultrasound (using sound waves) guidance to your affected shoulder. A repeat shoulder exam will be performed and recorded
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine
  Arms: Subacromial Lidocaine Injection
Drug: Saline
  Arms: Subacromial Saline Injection

SUMMARY:
Clinical manifestations of rotator cuff tear include shoulder pain, weakness, and stiffness. The level of pain is often a limiting factor when assessing shoulder range of motion and strength pre-operatively. Pain itself has even been a cause of weakness due to muscle atrophy.

The purpose of this study is to further understand the effect pain has by measuring constant shoulder scores in patients before and after ultrasound guided subacromial (the outer end of the shoulder blade) injection of lidocaine (a local anesthetic or numbing agent) compared to saline (salt solution), in patients indicated for arthroscopic rotator cuff repair. The saline and lidocaine has been approved for use by the U.S. Food and Drug Administration (FDA). The constant shoulder score includes your level of pain, activity level, range of motion and strength measures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is determined to have a full thickness rotator cuff tear (1-3 cm), on the pre-operative MRI scan or found arthroscopically, and is scheduled to undergo arthroscopic surgical repair
* Written informed consent is obtained

Exclusion Criteria:

* Revision Surgery
* Irreparable tear or partial tear
* Subscapularis involvement
* Any patient lacking decisional capability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Constant Shoulder Score | 10 minutes following injection
  Validated outcome score assessing pain and function of shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Brian Forsythe, MD, Principal Investigator — Rush University Medical Center

REFERENCES:
- [Derived] Forsythe B, Agarwalla A, Puzzitiello RN, Patel BH, Lu Y, Verma NN, Romeo AA, Cole BJ. Clinical Function Improves After Subacromial Injection of Local Anesthetic in Full-Thickness Rotator Cuff Tears: A Randomized Control Trial. Orthop J Sports Med. 2020 Jan 3;8(1):2325967119892331. doi: 10.1177/2325967119892331. eCollection 2020 Jan. PMID 31934594